CLINICAL TRIAL: NCT00547469
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Effectiveness of DDP733 in Female Patients With Irritable Bowel Syndrome With Constipation
Brief Title: A Study of the Safety and Effectiveness of DDP733 in Treating IBS With Constipation in Females
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dynogen Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DDP733-07-010
Record Dates: First submitted 2007-10-19; First posted 2007-10-22 (Estimated); Last update posted 2008-04-08 (Estimated); Status verified 2008-04

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; IBS-c; IBS constipation; women with IBS; women with constipation
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — DDP733

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: DDP733

SUMMARY:
This study will evaluate the safety and effectiveness of the investigational drug DDP733 in treating female patients with IBS-c. A placebo control will be utilized.

ELIGIBILITY:
Inclusion Criteria:

* Female from 18 to 65 years of age, inclusive
* Patient experiences recurrent abdominal pain or discomfort at least 3 days per month for the last 3 months with symptom onset at least 6 months prior to diagnosis. The patient's symptoms must be associated with 1 or more of the following:

  * Improvement with defecation
  * Onset associated with a change in frequency of stool
  * Onset associated with a change in form (appearance) of stool
* Negative serum and urine pregnancy tests
* Completion of at least six days of daily diary assessments using a phone-in information system prior to randomization

Exclusion Criteria:

* Serious underlying diseases, including psychiatric disorders
* Current history of conditions affecting bowel transit
* Recent history of biochemical or structural abnormalities of the gastrointestinal tract, gastrointestinal surgery, or gastrointestinal infection
* Clinically significant abnormal examination findings or laboratory tests
* Inability to stop taking certain medications, or a planned change in medications (including herbal remedies) which could interfere with study assessments
* Use of drugs and or ethanol which may interfere with compliance of study procedures or influence study outcome
* Presence of a medical condition which could interfere with the interpretation of study data
* Significant use of nicotine or caffeine

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2007-10

PRIMARY OUTCOMES:
Overall Subject Global Assessment (SGA) of relief of IBS symptoms, collected weekly

SECONDARY OUTCOMES:
Weekly assessments of abdominal discomfort/pain, bowel habit, and satisfaction with bowel habit.
Other secondary efficacy variables reflecting IBS symptoms include daily assessments of abdominal discomfort/pain; abdominal bloating, the number and consistency of stools, straining at defecation, and feeling of incomplete evacuation.

CONTACTS AND LOCATIONS:
Overall Officials: Dynogen Study Director, MD, Study Director — Dynogen Pharmaceuticals, Inc
Locations (69):
- United States (62):
  - Alliance Clinical Trials, Birmingham, Alabama
  - Clinical Research Associates, Huntsville, Alabama
  - Medical Affiliated Research Center, Inc., Huntsville, Alabama
  - Mobile Medical Diagnostic, Mobile, Alabama
  - Pivotal Research Centers, Peoria, Arizona
  - Genova Clinical Research, Tucson, Arizona
  - Arkansas Gastroenterology, Sherwood, Arkansas
  - Impact Clinical Trials, Beverly Hills, California
  - Discovery Clinical Research, Encinitas, California
  - Family Medical Center, Foothill Ranch, California
  - Digestive and Liver Disease Specialist, A Medical Group, Inc., Garden Grove, California
  - Prime Care Clinical Research, Inc., Mission Vejo, California
  - California Research Foundation, San Diego, California
  - Medical Center for clinical research, San Diego, California
  - Westlake Medical Research, Westlake Village, California
  - Clinical Trial Center of Colorado, LLC, Castle Rock, Colorado
  - Clinical Trials Management of Boca Raton, Inc., Boca Raton, Florida
  - Jupiter Research, Jupiter, Florida
  - AppleMed Research Inc., Miami, Florida
  - Accord Clinical Research, LLC, Port Orange, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Mount Vernon Clinical Research, Atlanta, Georgia
  - Atlanta Gastroenterology Associates, LLC, Marietta, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - Rosemark WomenCare Specialists, Idaho Falls, Idaho
  - Accelovance, Peoria, Illinois
  - Rockford Gastroenterology Associates, Ltd., Rockford, Illinois
  - Indiana Medical Research, LLC, Elkhart, Indiana
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Metropolitan Gastroenterology Group, PC Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Maryland Digestive Disease Research, LLC, Laurel, Maryland
  - Boston Clinical Trials, INC., Boston, Massachusetts
  - Women's Health Care Specialists, PC, Paw Paw, Michigan
  - CRC of Jackson, LLC at Jackson Medical Clinic, Jackson, Mississippi
  - Gastrointestinal Associates, P.A., Jackson, Mississippi
  - Center for Digestive and Liver Diseases, Inc., Mexico, Missouri
  - Lovelace Scientific Resources, Henderson, Nevada
  - LifeLine Research, Inc., Brooklyn, New York
  - UNC Center for Functional GI and Motility Disorders, Chapel Hill, North Carolina
  - Peters Medical Research dba Bethany Medical Center, High Point, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Piedmont Medical Research Associates, Winston-Salem, North Carolina
  - Hightop Medical Research Center, Cincinnati, Ohio
  - Gastroenterology Research Consultants of Greater Cincinnati, Cincinnati, Ohio
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Gastrointestinal and Liver Diseases Consultants, Dayton, Ohio
  - Clinical Trials Research Services, LLC, Pittsburgh, Pennsylvania
  - Southeastern Clinical Research, Chattanooga, Tennessee
  - Jackson Clinic, PA, Jackson, Tennessee
  - Regional Research Institute, Jackson, Tennessee
  - Gastroenterology Associates Clinical Research, Kingsport, Tennessee
  - Baylor College of Medicine, Baylor Clinic, Houston, Texas
  - DCOL Center for Research, Longview, Texas
  - Advanced Research Institute, Ogden, Utah
  - Virginia Mason Meidical Center, Seattle, Washington
  - Rowan Research, Spokane, Washington
  - Spokane Internal Medicine, Spokane, Washington
  - Wisconsin Center for Advanced Research Division of GI Associates, LLC, Milwaukee, Wisconsin
  - Aurora Health Center, Waukesha, Wisconsin
- Canada (7):
  - McMaster University Dept of Gastrointerology St. Joseph's Healthcare, Hamilton, Ontario
  - St. Joseph's Hospital, London, Ontario
  - Meadowlands Family Health Center, Ottawa, Ontario
  - London Road Diagnostic Clinic, Sarnia, Ontario
  - Sarnia Institute of Clinical Research, Sarnia, Ontario
  - Canadian Phase Onward Inc., Toronto, Ontario
  - Toronto Digestive Disease Associates, Inc., Toronto, Ontario